CLINICAL TRIAL: NCT02462135
Title: The Development and Evaluation of the Effectiveness of a Virtual Interactive Memory Training Program for Older Adults With Mild Cognitive Impairment: Protocol of a Randomized Controlled Study
Brief Title: Protocol of Virtual Interactive Memory-Training Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ministry of Science and Technology, Taiwan (Other Government)
Responsible Party: Principal Investigator, Yang, Hui-Ling, Ph.D. candidate, Ministry of Science and Technology, Taiwan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 201301045
Record Dates: First submitted 2015-05-28; First posted 2015-06-03 (Estimated); Last update posted 2017-12-15 (Actual); Status verified 2017-12

CONDITIONS: Mild Cognitive Impairment
Keywords: Mild cognitive impairment; Memory training; Randomized controlled study
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Cognitive Training

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Virtual interactive memory training (Experimental): Training sessions of the VIMT group are divided into initial training and booster training. Each training session is 45 minutes/day, 3 sessions/week, for 12 weeks for both initial training and booster training (36 sessions each).
  Interventions: Behavioral: Virtual interactive memory training
- Passive information activities (Active Comparator): The training of active control group is the same as VIMT group (45 min/day, 3 days/week, for 12 weeks, for a total of 36 sessions). The active control group receives only the initial training.
  Interventions: Behavioral: Passive information activities

INTERVENTIONS:
Behavioral: Virtual interactive memory training — Training sessions of the VIMT group are divided into initial training and booster training. Each training session is 45 minutes/day, 3 sessions/week, for 12 weeks for both initial training and booster training (36 sessions each). The training content of the four memory training include: (1) spatial encoding memory training task, (2) updating-spatial memory training task, (3) updating-visual memory training task, and (4) rehearsal-visuospatial memory training task.
  Other Names: Memory training
  Arms: Virtual interactive memory training
Behavioral: Passive information activities — The active control group (Passive information activities) only accepts the initial training phase, which training content of the two types to include: (1) listening to audio books, and (2) reading online newspaper.
  Other Names: Active control group
  Arms: Passive information activities

SUMMARY:
This study sought to investigate the changes in objective memory performance (including immediate recall and delayed recall), subjective memory complaints and degree of depression in older adults with mild cognitive impairment after Virtual interactive memory training (VIMT).

DETAILED DESCRIPTION:
This double-blind randomized controlled study has a 2-arm parallel group design. All subjects will be randomized by the block randomization, into intervention group (Virtual interactive memory training, VIMT), or active control group (Passive information activities, PIA). Training sessions of the VIMT group are 45 minutes/day, 3 days/week, for 12 weeks (36 sessions each). The training of PIA group is the same as VIMT group. We constructed a rigorous VIMT program adhering to the Consolidated Standards of Reporting Trials (CONSORT) reporting guidelines. The investigators expect to determine the improvement in memory function and degree of depression of older adults with mild cognitive impairment after using the VIMT.

ELIGIBILITY:
Inclusion Criteria:

1. Participants must endorse at least two items from a list of frequent subjective memory complaints by patient and/or an informant
2. Objective memory impairment on neuropsychological tests of memory 1.5 SD or more below age/education norms
3. Clinical neurologic examination by the Mini-Mental State Examination (MMSE) score of 24 or higher, and cut-off score of 23/24 on the Montreal Cognitive Assessment (MoCA)
4. No impairment in personal activities of daily living (P-ADL) as determined by clinical interview with participant and family

Exclusion Criteria:

1. The clinical diagnosis of dementia was based on the DSM-IV-TR
2. Active in another cognitive or memory-related training in the past year
3. Comorbid medical conditions that would predispose them to imminent functional decline or cognitive impairment
4. A diagnosis of major neurological or psychiatric illness history and/or behavioral problems that would sufficiently impair performance to make participation impossible
5. Severe losses in vision, hearing, or communicative ability

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-03; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Change in objective memory performance as measured by the Chinese version of the Wechsler Memory Scale-III (WMS-III). | Change from baseline in objective memory performance at Immediate post-test, 3 months, 6 months and one year after intervention.

SECONDARY OUTCOMES:
Change in subjective memory complaints as measured by the Multifactorial Memory Questionnaire (MMQ). | Change from baseline in subjective memory complaints at Immediate post-test, 3 months, 6 months and one year after intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Hui-Ling Yang, PhD, Principal Investigator — Taipei Medical University; Kuei-Ru Chou, Professor, Study Chair — Taipei Medical University
Locations (1):
- Residential care facilities, Taipei, Taiwan

REFERENCES:
- [Derived] Yang HL, Chu H, Kao CC, Chiu HL, Tseng IJ, Tseng P, Chou KR. Development and effectiveness of virtual interactive working memory training for older people with mild cognitive impairment: a single-blind randomised controlled trial. Age Ageing. 2019 Jul 1;48(4):519-525. doi: 10.1093/ageing/afz029. PMID 30989165